CLINICAL TRIAL: NCT05290454
Title: mNGS -Guided Antimicrobial Treatment Versus Conventional Antimicrobial Treatment in Early Severe Community-Acquired Pneumonia Among Immunocompromised Patients
Brief Title: mNGS -Guided Antimicrobial Treatment in Early Severe Community-Acquired Pneumonia Among Immunocompromised Patients
Acronym: MATESHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Wang Hao, associate professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wang Hao Qilu
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Severe Acute Respiratory Infection; Community-acquired Pneumonia; Respiratory Tract Infections; Pneumonia; Infections
Keywords: Metagenomic next generation sequencing; Community-acquired Pneumonia; Severe community acquired pneumonia; Conventional microbiology diagnosis technology; Antimicrobial therapy; Pneumonia; Respiratory Tract Infections
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Tract Infections; Pneumonia; Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mNGS-guided treatment group (Experimental): In mNGS-guided treatment group, participants undergo mNGS, using appropriate lower respiratory tract (LRT) specimen, and conventional microbiological diagnostic tests. LRT specimen, such as endotracheal aspiration (ETA), bronchoalveolar lavage fluid (BALF), or protected specimen brush (PSB), will be obtained within 24 hours after the participants entering the ICU. Conventional microbiology diagnostic techniques will be also applied using appropriate LRT specimens and other necessary specimens (such as blood, pleural fluid, urine, et al.). Clinicians alter or confirm the definitive treatment based on mNGS results, as well as results from conventional microbiology diagnostic techniques.
  Interventions: Other: mNGS-guided treatment
- Conventional treatment group (No Intervention): In conventional treatment group, participants undergo conventional microbiological tests using appropriate LRT specimen, and other necessary specimens (such as blood, pleural fluid, urine, et al.). LRT specimen, such as endotracheal aspiration (ETA), bronchoalveolar lavage fluid (BALF), or protected specimen brush (PSB), will be obtained within 24 hours after the participants entering the ICU. Based on results of conventional microbiology diagnostic techniques, clinicians alter or confirm the definitive treatment of participants.

INTERVENTIONS:
Other: mNGS-guided treatment — mNGS detect the causative microorganisms using appropriate lower respiratory tract (LRT) specimen. LRT specimen, such as endotracheal aspiration (ETA), bronchoalveolar lavage fluid (BALF), or protected specimen brush (PSB), will be obtained within 24 hours after the participants entering the ICU. Clinicians apply the definitive treatment based on mNGS results, as well as results of conventional microbiology diagnostic techniques.
  Arms: mNGS-guided treatment group

SUMMARY:
Severe Community-acquired pneumonia (SCAP) is a leading global infectious cause of intensive care unit (ICU) admission (approximately 20%-30%), and the primary reason of mortality and morbidity in immunocompromised patients. There is a global increase of patients with distinct immunocompromised conditions due to the advance of cancer treatment, increasing biologics, and immunosuppressants for autoimmune diseases and growing organ transplant recipients, and it has been estimated that patients with immunocompromised conditions account for approximately 35% of all intensive care unit (ICU) admissions. Immunocompromised patients with SCAP have more factors to complicate with sepsis, respiratory failure, acute respiratory distress syndrome, and the mortality rate can be up to 50%. With the aim to apply early accurate antimicrobial therapy to improve clinical prognosis of SCAP patients with immunocompromised conditions, timely identification of pathogen is particularly important. Conventional microbiological diagnostic methods such as standard microbiologic cultures, microscopy, polymerase chain reaction (PCR), respiratory virus multiplex PCR, as well as pathogen-specific antigens and antibody assays, are currently commonly used to detect pathogens, although they have various limitations. However, conventional antimicrobial therapy depends on the results of conventional diagnostic methods, which may delay timely accurate antimicrobial therapy at the initial stage, and the mortality of immunocompromised patients with SCAP may be increased. Metagenomic next-generation sequencing (mNGS), which can determine pathogens more quickly (usually within 24h) and accurately comparing with conventional diagnostic methods by analyzing cell-free nucleic acid fragments of pathogens using appropriate lower respiratory tract (LRT) specimen, is increasingly used in severe respiratory infectious disease, especially among immunocompromised patients. This study aims to determine whether mNGS (using LRT specimen) guided antimicrobial treatment improves clinical prognosis of SCAP patients with immunocompromised conditions when compared with conventional antimicrobial treatment.

DETAILED DESCRIPTION:
Severe Community-acquired pneumonia (SCAP) is an emergence infection disease of lung parenchyma that acquired outside of a hospital setting. SCAP is a leading global infectious cause of intensive care unit (ICU) admission (approximately 20%-30%), and the primary reason of mortality and morbidity in immunocompromised patients. There is a global increase of patients with distinct immunocompromised conditions due to the advance of cancer treatment, increasing biologics, and immunosuppressants for autoimmune diseases and growing organ transplant recipients, and it has been estimated that patients with immunocompromised conditions account for approximately 35% of all intensive care unit (ICU) admissions. Immunocompromised patients, who always at risk of mixed and unusual pathogens infection, have more factors to complicate with sepsis, respiratory failure, acute respiratory distress syndrome, and the mortality rate can be up to 50%. Moreover, the outcomes in immunocompromised patients with SCAP not only related to disease severity but also related to delays initiation of receiving appropriate therapy. 2019American Thoracic Society (ATS)/Infectious Diseases Society of America (IDSA) community-acquired pneumonia (CAP) guideline recommends that administering appropriate antimicrobials as soon as possible is the most effective measure to improve clinical prognosis and reduce mortality rate for SCAP patients. Therefore, timely identification of pathogenic microorganisms is particularly crucial for antimicrobial treatment in immunocompromised patients with SCAP.

Conventional microbiology diagnostic methods, such as standard microbiologic cultures, microscopy, polymerase chain reaction (PCR), respiratory virus multiplex PCR, as well as pathogen-specific antigens and antibody assays, are associated with relevant limitations: (1) long culture cycle and low positive rate; (2) usually only one pathogen can be detected at a time; (3) inability to detect fastidious or difficult culture organisms; (4) pathogen antibody-based testing may be unreliable in immunocompromised patients who are unable to mount antibody responses. Conventional diagnostic methods make big challenge for pathogens diagnosis of SCAP among immunocompromised patients due to above limitations and the complicated causative microorganisms. However, conventional antimicrobial therapy based on the results of conventional microbiology diagnostic techniques, which may delay timely accurate antimicrobial therapy at the initial stage, and the mortality of immunocompromised patients with SCAP may be increased. Metagenomic next-generation sequencing (mNGS), which can quickly (usually within 24h) detect a wide array of bacteria, viruses and fungi in an unbiased manner at the same time by analyzing cell-free nucleic acid (DNA) fragments of pathogens using appropriate lower respiratory tract (LRT) specimen, is increasingly used in severe infectious disease, especially among immunocompromised patients. This study speculates that mNGS (using LRT specimen) can guide early and accurate antimicrobial treatment for immunocompromised patients with SCAP. This multi-center, opening, randomized, controlled trail will enroll SCAP patients with immunocompromised conditions to determine whether mNGS-guided antimicrobial treatment improve the clinical prognosis and increase the clinical cure rate. The purpose of this study is to characterize the effect of mNGS-guided antimicrobial treatment for SCAP versus conventional treatment among immunocompromised patients. It is postulated that mNGS-guided antimicrobial treatment for immunocompromised patients with SCAP will improve clinical outcomes among these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of sever community acquired pneumonia (SCAP).

   SCAP is defined as:

   With either one major criterion or at least three minor criteria of the IDSA/ATS CAP severity criteria.
2. Admission in ICU.
3. Time from SCAP diagnosis to ICU admission<24 h.
4. Patients with Immunocompromised conditions.

Immunocompromised conditions are defined as:

1. Use of long-term (>3 months) or high-dose (>0.5 mg/kg/d) steroids.
2. Use of other immunosuppressant drugs.
3. Solid organ transplantation.
4. Solid tumor requiring chemotherapy in the last 5 years.
5. Hematologic malignancy regardless of time since diagnosis and received treatments.
6. Primary immune deficiency.
7. HIV infection with a cluster of differentiation 4 (CD 4) T-lymphocyte count <200 cells/ml or percentage <14%.
8. Laboratory tests show absolute neutrophil count < 1,000 cells/µl on ICU admission.
9. Other immunosuppression status judged by the physicians.

Exclusion Criteria:

1. Age<18 years old.
2. Pregnant or lactating women.
3. Those who are expected to die within 72 h.
4. Receiving palliative therapy or supportive treatment only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The relative change in Sequential Organ Failure Assessment (SOFA) score from randomization to day 5, day 7, day 10, or the day of ICU discharge/death | at day 5, day 7,and day 10 after randomization or the day of ICU discharge/death
  Relative Changes in sequential organ failure assessment (SOFA) score at day 5,day 7 and day 10,or the day of ICU discharge/death after randomization when compared with day 0. Sequential organ failure assessment (SOFA) score is used to describe quantitatively and as objectively as possible the degree of organ dysfunction/failure over time. We will record the worst value from randomization until day 10 or the day of ICU discharge/death. The score value is among 0-24, and the higher score value means the worse outcome.
the consumption of antimicrobial agents during ICU stay (expressed as defined daily doses) | at 28-day and 90-day after randomization
  The consumption of antimicrobial agent during participants' ICU stay, and the consumption will be calculated by in terms of defined daily doses (DDD) available from the World Health Organization (WHO).

SECONDARY OUTCOMES:
days from randomization to initiation of definitive antimicrobial treatment | during 28 days after randomization
  The duration from SCAP diagnosis to the first dose of appropriate definitive antibiotic usage.
overall antimicrobial agent use and cost | at 28-day and 90-day after randomization
  The consumption and cost of antimicrobial agent from admission to discharge of hospital or death
length of ICU stay | at 28-day and 90-day after randomization
  The duration from admission to discharge of ICU or death.
28- and 90-day all-cause mortality | at 28-day and 90-day after randomization
  Mortality at 28- and 90-day after randomization.
Clinical cure rate | at 28-day and 90-day after randomization
  Clinical cure is defined as resolution of clinical signs and symptoms, and no requirement for continue antimicrobial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Hao associate professor, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form will be shared with other researchers when start this trial.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and ICF will be shared with other researchers when start this trial for five years.
Access Criteria: Ever researchers can access our study protocol and ICF from the web of clinical trials.gov.

REFERENCES:
- [Derived] Fan S, Si M, Xu N, Yan M, Pang M, Liu G, Gong J, Wang H. Metagenomic next-generation sequencing-guided antimicrobial treatment versus conventional antimicrobial treatment in early severe community-acquired pneumonia among immunocompromised patients (MATESHIP): A study protocol. Front Microbiol. 2022 Aug 2;13:927842. doi: 10.3389/fmicb.2022.927842. eCollection 2022. PMID 35983331

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT05290454/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05290454/ICF_001.pdf